CLINICAL TRIAL: NCT00957593
Title: Induction of Labor With Oxytocin: When Should Oxytocin be Held?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Joanne Quinones, MD, Attending Physician, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-20080907
Record Dates: First submitted 2009-07-31; First posted 2009-08-12 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Labor Induction; Cesarean Delivery
Keywords: Induction of labor in term pregnancies; Term pregnancy; Cesarean delivery
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Active Comparator): Continuation of oxytocin per protocol once the patient reaches active labor
  Interventions: Drug: Oxytocin
- Oxytocin discontinuation (Active Comparator): Oxytocin will be stopped once the patient reaches active labor
  Interventions: Drug: Oxytocin discontinuation

INTERVENTIONS:
Drug: Oxytocin — Continuation of oxytocin once in active labor
  Arms: Oxytocin
Drug: Oxytocin discontinuation — Oxytocin will be stopped once in active labor
  Arms: Oxytocin discontinuation

SUMMARY:
The investigators propose to perform a prospective randomized control trial to compare the rate of cesarean delivery in women where Oxytocin (OT) is discontinued once active labor begins (5 cm dilation) when compared with women where OT is continued at a maintenance level per the usual protocol.

One study group will follow an oxytocin protocol which is incremental until 5 cm dilation and then maintained at the same level throughout labor. The second arm will follow an oxytocin protocol also incremental, but then discontinued once the cervix is 5 cm. The primary outcome will be the rate of cesarean delivery between the groups. Secondary outcomes to be evaluated will include duration of the labor, fetal heart rate abnormalities, and frequency of uterine hyperstimulation, maternal and neonatal outcomes.

As mentioned in the study proposal, the proposed experimental arm is currently not performed as part of the oxytocin guidelines at the investigators' institution. One study from Israel suggests no difference in pregnancy outcomes with the proposed use of oxytocin. Although some providers stop the oxytocin in active labor for their patients, this is not a commonly performed procedure at the investigators' institution. The investigators are not aware of other institutions employing the above practice.

DETAILED DESCRIPTION:
Oxytocin is the most common agent used to induce and augment labor. Oxytocin injection is approved by the Food and Drug Administration for the initiation or improvement of uterine contractions to achieve vaginal delivery. It is used to induce labor and stimulate or reinforce labor.

The relationship of oxytocin and its receptor is crucial in obtaining adequate uterine activity and thus inducing active labor. Due to this very balanced relationship, a question exists about the optimal regimen of oxytocin administration for induction of labor and on how long to continue oxytocin once active labor begins. Some literature suggests that once in the active phase of labor oxytocin may be discontinued without altering the progression of labor. The objective of this study is to determine whether there is an increased rate of cesarean delivery in women undergoing induction of labor when oxytocin is discontinued in the active phase of labor.

Blair-Bell was the first who, in 1909, demonstrated the uterotonic action of posterior pituitary extracts at a cesarean delivery. Since then oxytocin, synthesized by du Vigneaud et al, has been most commonly used for the induction of labor. Oxytocin (OT) is a polypeptide hormone, synthesized in the hypothalamus and in reproductive tissues during pregnancy.

Oxytocin stimulates uterine contraction by mechanisms involving the activation of receptor-operated calcium channels. Calcium-dependent phosphorylation of myosin triggers the interaction of myosin and actin subunits throughout the uterus leading to contractions.

During labor and parturition the relationship between oxytocin and its receptor is critical in achieving adequate uterine contractions and thus active labor. If few receptors are present, as seen in an early gestation, a large amount of OT is required for contractions. The opposite is true in term pregnancy. OT binding to its receptor is very important because excess doses of OT are not productive and may have undesirable effects.

The use of OT can cause hyperstimulation (excessive contractions leading to abnormal fetal heart rate patterns) even when used in adequate doses. Nonetheless, induction of labor with OT can be beneficial in reducing the incidence of prolonged labor and subsequent cesarean delivery without increasing perinatal morbidity or mortality.

Currently OT protocols vary throughout hospitals. Both low and high dose regimens as outlined by the American College of Obstetrician and Gynecologists are appropriate for labor induction. At our facility intravenous OT is started at 1-2 milliunits per minute and increased by 2 milliunits every 15 minutes until obtaining normal progression of labor usually at 150-300 Montevideo units on the contraction monitor. Low dose regimens with less frequent increases in dose are associated with decreased hyperstimulation. However use of high-dose oxytocin has not been found to increase the incidence of birth asphyxia or perinatal morbidity.

As mentioned in the study proposal, the proposed experimental arm is currently not performed as patient of the oxytocin guidelines at our institution. One study from Israel found no difference in pregnancy outcomes with the proposed use of oxytocin. Although we are aware of one provider that stops the oxytocin drip once the patient is in active labor, this is not a commonly performed procedure at our institution. We are not aware of other institutions employing the above.

We propose to perform a prospective randomized control trial to compare the rate of cesarean delivery in women where OT is discontinued once active labor begins (5 cm dilation) when compared with women where OT is continued at a maintenance level per the usual protocol.

One study group will follow an oxytocin protocol which is incremental until 5 cm dilation and then maintained at the same level throughout labor. The second arm will follow an oxytocin protocol also incremental, but then discontinued once the cervix is 5cm. The primary outcome will be the rate of cesarean delivery between the groups. Groups will be stratified by parity (nulliparous vs. multiparous). Secondary outcomes to be evaluated will include duration of the labor, fetal heart rate abnormalities, and frequency of uterine hyperstimulation, maternal and neonatal outcomes.

Based on our sample size calculation, we will need at least 160 patients in each arm of the study to find an increase in the cesarean delivery rate from 25% to 40% in women who undergo induction of labor where oxytocin is discontinued once the active phase of labor begins. This sample size calculation uses a power of 80% and an alpha level (statistical significance) of 0.05. The baseline rate of cesarean in the US is 25-30%. We chose 40% as a significantly increased rate of CS since this rate would represent a 60% increase in CS from the baseline risk in the population.

We are looking for a difference in cesarean rates between the experimental arm and the maintenance arm. Evaluating the data as an equivalence study (no difference between the interventions) would significantly increase the sample size needed for the study. With our current sample size calculation, if a cesarean rate difference is not found between the groups (meaning discontinuation of oxytocin is not inferior to the maintenance use of oxytocin in active labor), we can state that our data do not support a significant increase (60% increase) in the risk of cesarean delivery rate when reducing the amount of oxytocin used for induction of labor.

It is not possible to blind the providers, nurses or patients to the arm of the study since oxytocin infusions need to be titrated and dosing level is important in managing labor. This will be an intention to treat analysis.

The decision to perform a cesarean delivery will be according to standard obstetric indications and will be ultimately decided by the treating physician, regardless of treatment assignment. Obstetric criteria are in place to perform cesarean deliveries. The treating physician at any time may restart the oxytocin in patients originally assigned to the oxytocin discontinuation arm.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for the study are pregnant women (with one fetus) scheduled for induction of labor with oxytocin at term gestation or greater, regardless of the indication for induction, bishop score (cervical dilation) or parity.

Exclusion Criteria:

* Exclusions include women with multiple gestations, previous cesarean sections, and documented fetal anomalies.
* Women with contraindications to labor or induction will also be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne N Quinones, MD MSCE, Principal Investigator — Lehigh Valley Health Network
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

REFERENCES:
- [Result] Diven LC, Rochon ML, Gogle J, Eid S, Smulian JC, Quinones JN. Oxytocin discontinuation during active labor in women who undergo labor induction. Am J Obstet Gynecol. 2012 Dec;207(6):471.e1-8. doi: 10.1016/j.ajog.2012.08.035. Epub 2012 Sep 7. PMID 22989707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ROUTINE oxytocin 127 Discontinuation of oxytocin 125
Period: Overall Study
Arm/Group | Oxytocin | Oxytocin Discontinuation
Started | 127 | 125
Completed | 127 | 125
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Oxytocin Discontinuation | Total
Number analyzed (Participants) | 127 | 125 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 125 | 252
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.6) | 27.7 (5.7) | 27.4 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 125 | 252
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 125 | 252

OUTCOME MEASURES:

1. Primary Outcome: Cesarean Delivery
Description: Mode of delivery is the primary outcome
Time Frame: 24-72 hours from admission for induction
Measure: Number; unit: Cesarean deliveries
Arm/Group | Oxytocin | Oxytocin Discontinuation
Number analyzed (Participants) | 127 | 125
Cesarean deliveries | 32 | 24

2. Secondary Outcome: Perinatal Outcomes
Description: Perinatal outcomes for patients included in the randomized trial
Time Frame: 24-72 hours
Population: Routine use of oxytocin vs discontinuation of oxytocin once in active labor 127 ROUTINE 125 discontinuation
Measure: Count of Participants; unit: Participants
Groups:
- Routine: Routine use of oxytocin vs discontinuation of oxytocin once in active labor
- Discontinuation: Oxytocin discontinued in the active phase of labor
Arm/Group | Routine | Discontinuation
Number analyzed (Participants) | 127 | 125
Participants
  Male gender | 70 | 66
  Neonatal resuscitation | 9 | 7
  Admission to NICU | 10 | 9
  Neonatal antibiotic use | 9 | 16

ADVERSE EVENTS:
Time Frame: Period for which data were collected includes the duration of the study, February 2009 to August 2011.
Groups:
- Oxytocin Arm: no adverse effects noted amongst the 252 patients enrolled in the study 127 in ROUTINE 125 in DISCONTINUATION ARM
- Oxytocin Discontinuation: Oxytocin discontinuation in the active phase of labor
Arm/Group | Oxytocin Arm | Oxytocin Discontinuation
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/125
Other Adverse Events (participants affected / at risk) | 0/127 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes